CLINICAL TRIAL: NCT07143773
Title: SGLT2i Safety and Efficacy on Kidney Allograft Function in Non-diabetic Kidney Transplant Recipients: A Randomized, Double-blind, Placebo Controlled, National, Multicenter Trial
Brief Title: SGLT2i Safety and Efficacy on Kidney Allograft Function in Non-diabetic Kidney Transplant Recipients
Acronym: SGL-TX-GFR
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Aarhus University Hospital (Other); Copenhagen University Hospital, Denmark (Other); Gødstrup Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EU CT:2024-518773-33-00
Record Dates: First submitted 2025-07-30; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-07

CONDITIONS: Kidney Transplantation Recipients; Sodium-Glucose Transporter 2 Inhibitors; Non-Diabetic Patients; Randomized Controlled Trial; Placebo Control Design
Keywords: SGLT2i; Kidney Transplant; Kidney Transplant Recipients; non-diabetic patients; Sodium-glucose Transporter 2 inhibitors; RCT
MeSH Terms: interventions — Sodium-Glucose Transporter 2 Inhibitors

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, placebo controlled, national, multicenter trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SGLT2i (Active Comparator): Daily dose of SGLT2i (Forxiga 10 mg tablet)
  Interventions: Drug: SGLT-2 inhibitor
- Placebo (Placebo Comparator): Daily dose of placebo tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SGLT-2 inhibitor — The intervention in this clinical trial will be treatment with an SGLT2 inhibitor (Forxiga, 10 mg tablet once daily) compared with a matching placebo. A total of 88 non-diabetic kidney transplant recipients will be enrolled. All participants will be randomized in a 1:1 ratio to receive either Forxiga or placebo as an add-on to standard immunosuppressive therapy. This intervention differs from other studies by specifically targeting non-diabetic kidney transplant recipients, a population in which the efficacy and safety of SGLT2 inhibitors have not yet been established.
  Arms: SGLT2i
Drug: Placebo — The control intervention in this clinical trial will be a matching placebo tablet, identical in appearance to Forxiga (10 mg), administered once daily as an add-on to standard immunosuppressive therapy. A total of 88 non-diabetic kidney transplant recipients will be enrolled. All participants will be randomized in a 1:1 ratio to receive either placebo or Forxiga. This placebo intervention ensures blinding of both participants and investigators and allows a direct comparison of the safety and efficacy of SGLT2 inhibition versus no active treatment in this unique patient population.
  Arms: Placebo

SUMMARY:
This clinical trial investigates whether 18 months of daily SGLT2i (10 mg Forxiga) preserves kidney function and evaluates safety, based on eGFR changes and adverse event occurrence in non-diabetic kidney transplant recipients.

The main questions it aims to answer are:

* Does SGLT2i versus placebo, as an add-on to standard care, preserve kidney transplant function in non-diabetic recipients?
* Is SGLT2i treatment safe for non-diabetic transplant recipients when evaluating adverse events?
* Does SGLT2i versus placebo affect the occurrence of urinary tract infections, post-transplant diabetes mellitus (PTDM) and prediabetes incidence, U-ACR, as well as renal and cardiovascular parameters?

Researchers will compare a daily dose of SGLT2i (10 mg Forxiga) with a placebo (a look-alike tablet with no active medicine).

Kidney transplant recipients who do not have diabetes can take part if they meet the study's requirements. Participants will be randomly assigned to receive either Forxiga or placebo once daily for 18 months. All participants will have check-ups every 3 months, which will include urine tests and blood samples. Neither the participants nor the study doctors will know which treatment they are receiving.

DETAILED DESCRIPTION:
Background:

Kidney transplantation is the best treatment for end-stage renal disease (ESRD), although the median allograft survival is only 15 years. In non-transplant patients with chronic kidney disease (CKD), sodium-glucose co-transporter type 2 inhibitors (SGLT2i) protect kidney function and slow the decline in estimated glomerular filtration rate (eGFR).

With the current kidney transplant survival of approximately 15 years, about one in ten adult kidney transplant recipients (KTR) outlive their donated kidneys. This poses a significant burden on both patients and society, increasing the demand for new transplantations. WHO reported a 9% increase in the number of kidney transplant recipients from 2022 to 2023. Therefore, research aimed at extending the functional lifespan of kidney transplants is crucial.

The efficacy of SGLT2i in KTR remains untested, and safety concerns persist, particularly regarding their impact on kidney transplant function. This study aims to investigate the safety and efficacy of this new class of anti-diabetic drugs (SGLT2i) on kidney transplant function. In the long-term, the investigators hope to contribute knowledge that will help preserve kidney transplant function, benefit society, and improve patients' quality of life.

Hypothesis:

The research team hypothesize that SGLT2i will not worsen kidney transplant function (eGFR) in non-diabetic KTR as an add-on to standard-of-care.

Research Objective:

In this non-inferior randomized controlled clinical trial the investigators will determine the safety and efficacy of oral SGLT2i compared with placebo as add-on to standard-of-care on effecting kidney transplant function in non-diabetic KTR.

The secondary objectives will evaluate the effect of oral SGLT2i compared with placebo as add-on to standard-of-care on urinary tract infection, incidence of PTDM and prediabetes status, U-ACR, renal parameters, cardiovascular parameters and adverse events in non-diabetic KTR.

The tertiary objective will be to evaluate the patients' overall health assessment using the SF-36 questionnaire.

Study Design:

An investigator-initiated, placebo-controlled, double-blinded, parallel-group, randomized, national, multicenter intervention study.

Methods:

Non-diabetic KTRs who are more than 6 months post kidney transplant will be randomized 1:1 to receive either 18 months of oral SGLT2i treatment (Forxiga 10 mg once daily) or placebo, both as add-ons to standard immunosuppressive therapy. Participants will have follow-ups after one week, four weeks, and then every 3 months for the remainder of the trial period. Each participant will be monitored through blood and urine laboratory tests, with efficacy and safety assessed at every visit by a nephrologist. Kidney transplant function will be estimated by ΔeGFR.

Blood and urine samples will be collected through the hospital laboratories entirely on an outpatient basis, as patients are accustomed to, 1-7 days prior to planned telephone or in-person follow-up appointments.

Primary endpoint:

- Kidney transplant function, determined by the chronic eGFR slope (ml/min/1.73m²), measured from week 4 and every 3 months thereafter until 18 months post-randomization.

Secondary endpoints:

* Acute eGFR slope (ml/min/1.73m²): Measured from baseline until week 4.
* Urine albumin/creatinine ratio (U-ACR) (mg/g).
* Blood parameters: Creatinine (µmol/L), Total cholesterol, LDL and HDL cholesterol, Triglycerides, Tacrolimus concentration (µg/L, clinical routine), ALAT (U/L), Bilirubin, Pro-BNP, Renin, angiotensin-2, and aldosterone.
* Urinary tract infection: Positive culture.
* Incidence of PTDM and prediabetes status by HbA1c (mmol/mol), random blood glucose (mmol/L) and Continuous glucose monitoring: Dexcom G7 Pro sensor, 10 days at visit 5 (3 months post-randomization).
* Change in volume status: Week 1 of therapy (weight).
* Incidence of kidney transplant rejection: Biopsy-verified.
* Renal composite outcome: Incidence of graft failure (defined as return to dialysis or retransplantation), Incidence of ESRD (eGFR < 15 ml/min/1.73m²), Incidence of > 25% increase in creatinine.
* Change in blood pressure: Systolic (SysBP, mmHg) and diastolic (DiaBP, mmHg).
* Relative incidence of out-of-target clinical routine blood Tacrolimus levels.
* Urine biomarkers: Indicators of podocyte and tubular function from selected sites.

Incidence of:

* Adverse events,
* Serious adverse events,
* Serious adverse reactions,
* All-cause mortality,
* Major Adverse Cardiac Events (MACE):

  * Death from cardiovascular causes,
  * Nonfatal myocardial infarction (AMI), including both STEMI and NSTEMI (ICD-10 codes):

    * I21.0 - Acute transmural myocardial infarction of the anterior wall,
    * I21.1 - Acute transmural myocardial infarction of the posterior wall,
    * I21.2 - Acute transmural myocardial infarction of other localization,
    * I21.3 - Acute subendocardial myocardial infarction,
    * I21.4 - Acute myocardial infarction without ST-elevation (NSTEMI),
    * I21.9 - Acute myocardial infarction, unspecified,
    * Reinfarction and complications of AMI:

      * I22.0-I22.9 - Reinfarction (a new AMI within 28 days after a previous AMI),
      * I23.0-I23.9 - Complications following acute myocardial infarction (e.g., papillary muscle rupture, ventricular septal defect, pericardial effusion).
  * Therapeutic coronary procedures: Coronary-artery bypass graft, percutaneous transluminal coronary angioplasty, or stenting,
  * Heart failure: Reduced ejection fraction (HFrEF) < 40%,
  * Nonfatal ischemic stroke: Diagnosed by CT or MRI of the brain,
  * Nonfatal haemorrhagic stroke: Diagnosed by CT or MRI of the brain,
  * Carotid procedures: Endarterectomy or stenting,
  * All vascular interventions: Revascularization, percutaneous transluminal angioplasty, or stenting
  * Peripheral limb amputation.

Tertiary endpoint:

- SF-36 (Short Form Health Survey 36)

Study population:

88 non-diabetic KTRs, more than 6 months post-transplant and with an eGFR > 25 ml/min/1.73m², will be recruited from the kidney transplant outpatient clinics at Odense University Hospital (OUH), Aarhus University Hospital (AUH), Rigshospitalet (RH), and Regionshospitalet Gødstrup (RHG) in Denmark. Participants will be randomized to receive either SGLT2i or placebo treatment for a minimum of 18 months after providing signed informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Obtained written informed consent
* Male or female patients, age ≥ 18 years.
* Non-diabetic KTR
* > 6 months post-transplant
* eGFR> 25 ml/min/1.73m2 within the last 3 months pre randomization
* Immunosuppressive must include Tacrolimus
* Negative plasma hCG in fertile women*, and acceptance of the use of contraception during the course of the study.

Exclusion Criteria:

* Patients treated (diet or antidiabetics) for diabetes type 1 or 2 before randomization
* eGFR< 25 ml/min/1.73m2 (before randomization)
* Alanine aminotransferase (ALAT) > 3 x upper normal limit
* Bilirubin > 2 x upper normal limit
* Pregnancy
* Breastfeeding
* Known allergy towards SGLT2i or the content substance
* Known intestinal bowel disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Kidney transplant function | Measured from week 4, and then every 3. month until 18. month post randomization.
  Chronic eGFR slope (ml/min/1.73m2)

SECONDARY OUTCOMES:
Incidence of PTDM and prediabetes status | Measured from week 4, and then every 3. month until 18. month post randomization.
  Evaluated by
  * HbA1c (mmol/mol)
  * Random blood glucose (mmol/L)
  * Continuous glucose monitoring with a Dexcom G7 pro sensor, 10 days on visit 5 (3 months post randomization)

OTHER OUTCOMES:
Proteinuria | Measured from week 4, and then every 3 month until 18 month post randomization.
  Urine albumin/creatinine ratio (U-ACR) (mg/g)

CONTACTS AND LOCATIONS:
Overall Officials: Lotte B Lange, MD, Principal Investigator — Department of Nephrology, Odense University Hospital
Locations (1):
- Department of Nephrology, Odense University Hospital Kløvervænget 6, Enterance 93, 2. floor, Odense, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data Available:
  Individual participant data (IPD) that underlie the results reported in the published article will be shared after de-identification. This includes text, tables, figures, and appendices.
  Supporting Documents:
  The study protocol and statistical analysis plan will also be made available.
  Time Frame:
  Data will be shared immediately following publication. There is no specified end date for availability.
  Criteria for Access:
  Data will be shared with researchers who submit a methodologically sound proposal aimed at achieving the goals outlined in their approved research proposal.
  Access Mechanism:
  Interested researchers should direct their proposals to:
  lotte.borg.lange@rsyd.dk. To gain access, requestors will be required to sign a data access agreement.
  Data Storage:
  The data will be stored for 25 years on a secure third-party platform (OPEN).
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The data will be available after the last patients last visit, which is estimated for summer 2027
  Data Storage:
  The data will be stored for 25 years on a secure third-party platform (OPEN).
Access Criteria: Criteria for Access:
  Data will be shared with researchers who submit a methodologically sound proposal aimed at achieving the goals outlined in their approved research proposal.
  Access Mechanism:
  Interested researchers should direct their proposals to:
  lotte.borg.lange@rsyd.dk. To gain access, requestors will be required to sign a data access agreement.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-05-15): https://cdn.clinicaltrials.gov/large-docs/73/NCT07143773/Prot_SAP_000.pdf